CLINICAL TRIAL: NCT03541213
Title: Impact de la Carence Martiale et de Son Traitement Sur le métabolisme Mitochondrial du Cardiomyocyte (MitoCardioFer)
Brief Title: Impact of Iron Deficiency and Its Correction on Mitochondrial Metabolism of the Cardiomyocyte (MitoCardioFer)
Acronym: MitoCardioFer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Angers (Other Government)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 2017-A00904-49
Record Dates: First submitted 2018-05-17; First posted 2018-05-30 (Actual); Last update posted 2022-07-29 (Actual); Status verified 2022-07

CONDITIONS: Iron-deficiency; Valvular Heart Disease
Keywords: ferric carboxymaltose; mitochondrial metabolism; cardiomyocyte
MeSH Terms: conditions — Anemia, Iron-Deficiency; Heart Valve Diseases | interventions — Blood Specimen Collection

STUDY DESIGN:
Intervention Model Description: 3 groups will be performed depending on the presence or absence of a pre-operative iron deficiency and whether they had an iron treatment preoperatively (before their inclusion in the study). However, patient management will not be different in the different groups from their inclusion in the study. Therefore we can consider that there is a single interventional group.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control group (Other): Patients with no iron deficiency prior to inclusion and who did not receive intravenous iron prior to inclusion.
  Intervention : myocardial biopsy, sternal bone marrow biopsy and blood sample (as in the other arms)
  Interventions: Procedure: myocardial biopsy; Procedure: sternal bone marrow biopsy; Biological: blood sample
- Iron deficiency group (Other): Patients with iron deficiency who did not receive intravenous iron prior to inclusion.
  Intervention : myocardial biopsy, sternal bone marrow biopsy and blood sample (as in the other arms)
  Interventions: Procedure: myocardial biopsy; Procedure: sternal bone marrow biopsy; Biological: blood sample
- Iron treated group (Other): Patients with iron deficiency who received intravenous iron prior to inclusion (greater than or equal to 1 g ferric carboxymaltose).
  Intervention : myocardial biopsy, sternal bone marrow biopsy and blood sample (as in the other arms)
  Interventions: Procedure: myocardial biopsy; Procedure: sternal bone marrow biopsy; Biological: blood sample

INTERVENTIONS:
Procedure: myocardial biopsy — Myocardial biopsy (after opening cardiac cavities under general anesthesia for valvular surgery) for mitochondrial metabolism analyses.
Procedure: sternal bone marrow biopsy — Sternal bone marrow biopsy (after sternal opening under general anesthesia for valvular surgery) for the quantification of iron stores
Biological: blood sample — blood sample (under general anesthesia for valvular surgery, using the arterial catheter already in place) for hepcidin quantification (hormone not dosed in the usual martial assessment)

SUMMARY:
Iron is involved in essential functions of the body. It allows the transport of oxygen in the blood, via hemoglobin, at the muscular level, via myoglobin, and it is also involved in cellular metabolism in general, in particular for the production of ATP at the mitochondrial level, within the cytochromes and iron-sulfur proteins of the respiratory chain.

Recently, iron deficiency has been identified as an important prognostic factor in heart failure patients. Iron therapy improves symptoms and physical performances of heart failure patients, even in the absence of anemia. As a result, the correction of iron deficiency is now proposed as one of the therapies for heart failure. However, the pathophysiology of the association between cardiac dysfunction and iron deficiency is still poorly understood.

The investigators previously developed a mouse model of iron deficiency without anemia, in which the investigators observed impaired physical performances, a decrease of left ventricular ejection fraction, and a decrease in mitochondrial complex I activity. These abnormalities were normalized after iron injection. These animal data suggest that iron deficiency is responsible for left ventricular dysfunction secondary to mitochondrial I complex abnormalities, and that iron therapy corrects them.

Iron deficiency is very common in the preoperative period of cardiac surgery, affecting 40 to 50% of patients. During this surgery, it is possible to perform a myocardial biopsy without risk to the patient.

The purpose of this study is to verify in patients requiring valvular heart surgery, if iron deficiency is responsible for a decrease in mitochondrial complex I activity and a decrease in cardiac function during the perioperative period, and to verify whether iron treatment improves these abnormalities.

DETAILED DESCRIPTION:
Iron is involved in essential functions of the body. It allows the transport of oxygen in the blood, via hemoglobin, at the muscular level, via myoglobin, and it is also involved in cellular metabolism in general, in particular for the production of ATP at the mitochondrial level, within the cytochromes and iron-sulfur proteins of the respiratory chain.

Iron deficiency has been shown to be responsible for fatigue and muscle weakness, regardless of the presence of an anemia. Recently, iron deficiency has been identified as an important prognostic factor in heart failure patients, with a prevalence increasing with NYHA class level, and association with mortality. Iron therapy improves the symptoms of heart failure patients and the 6-minute walk test, even in the absence of anemia. The correction of iron deficiency is now proposed as one of the therapies for heart failure. However, the pathophysiology of the association between cardiac dysfunction and iron deficiency is still poorly understood.

The investigators previously developed a mouse model of iron deficiency without anemia, in which the investigators observed impaired physical performances, a decrease of left ventricular ejection fraction, and a decrease in mitochondrial complex I activity. These abnormalities were normalized after iron injection. These animal data suggest that iron deficiency is responsible for left ventricular dysfunction secondary to mitochondrial I complex abnormalities, and that iron therapy corrects them.

Iron deficiency is very common in the preoperative period of cardiac surgery, affecting 40 to 50% of patients. During this surgery, it is possible to perform a myocardial biopsy without risk to the patient. There is therefore an opportunity to further explore the impact of iron deficiency and its treatment on mitochondrial energy metabolism of cardiomyocytes. We hypothesize that the activity of the mitochondrial complex I is decreased in the presence of iron deficiency and that the iron treatment corrects this decrease.

The purpose of this study is to verify in patients requiring valvular heart surgery, if iron deficiency is responsible for a decrease in mitochondrial complex I activity and a decrease in cardiac function during the perioperative period, and to verify whether iron treatment improves these abnormalities.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Patients that must be operated for a valvular heart surgery (aortic or mitral) scheduled in the month which follows the anaesthesia consultation (visit of inclusion)
* The preoperative iron status is known
* Patient signed informed consent

Exclusion Criteria:

* Refusal of the patient to participate
* Refusal of the surgeon or the anaesthetist who are responsible of patient management
* Patients with a known iron overload (for example : hemochromatosis)
* Counter-indication in the realization of a sternal bone marrow biopsy or myocardial biopsy (for example : endocarditis)
* Adult patients under legal guardianship
* Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 55 (Actual)
Dates: Start 2019-01-23 (Actual); Primary Completion 2020-09-07 (Actual); Study Completion 2020-09-07 (Actual)

PRIMARY OUTCOMES:
Measure of the maximal activity of the mitochondrial complex I using spectrometry | At the time of the myocardial biopsy
  Measure of the maximal complex I activity using spectrometry on isolated mitochondria from myocardial biopsy.

SECONDARY OUTCOMES:
Measure of the maximal activity of the others mitochondrial complexes using spectrometry (Complexes II, III and IV) | At the time of the myocardial biopsy
Quantification of the number of mitochondria per cardiomyocyte using Western-Blot | At the time of the myocardial biopsy
Quantification and analysis of the complex I assemblage using BN-PAGE | At the time of the myocardial biopsy
Quantification of myoglobin in cardiomyocytes using Western-Blot | At the time of the myocardial biopsy
Cardiac function using echocardiography in pre-, intra- and post-operative periods | At the time of the myocardial biopsy

CONTACTS AND LOCATIONS:
Overall Officials: RINEAU Emmanuel, MD, Principal Investigator — University Hospital
Locations (1):
- CHU Angers - DEPARTEMENT D'ANESTHESIE REANIMATION, Angers, France